CLINICAL TRIAL: NCT01763918
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate Safety, Tolerability and Efficacy of AMG 145 on LDL-C in Subjects With Heterozygous Familial Hypercholesterolemia
Brief Title: Reduction of LDL-C With PCSK9 Inhibition in Heterozygous Familial Hypercholesterolemia Disorder Study-2
Acronym: RUTHERFORD-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20110117; 2012-001365-32 (EudraCT Number)
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Hyperlipidemia
Keywords: High cholesterol, Treatment for high cholesterol, Lowering cholesterol, Lowering high cholesterol, Hypercholesterolemia
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo Q2W (Placebo Comparator): Participants received placebo subcutaneous injection once every 2 weeks (Q2W) for up to 12 weeks.
  Interventions: Drug: Placebo
- Placebo QM (Placebo Comparator): Participants received placebo subcutaneous injection once every month (QM) for up to 12 weeks.
  Interventions: Drug: Placebo
- Evolocumab Q2W (Experimental): Participants received 140 mg evolocumab by subcutaneous injection once every 2 weeks for up to 12 weeks.
  Interventions: Biological: Evolocumab
- Evolocumab QM (Experimental): Participants received 420 mg evolocumab by subcutaneous injection once a month for up to 12 weeks.
  Interventions: Biological: Evolocumab

INTERVENTIONS:
Biological: Evolocumab — Administered by subcutaneous injection
  Other Names: AMG 145; Repatha
  Arms: Evolocumab Q2W; Evolocumab QM
Drug: Placebo — Administered by subcutaneous injection
  Arms: Placebo Q2W; Placebo QM

SUMMARY:
The primary objective was to evaluate the effect of 12 weeks of evolocumab subcutaneously once every 2 weeks (Q2W) and once monthly (QM), compared with placebo, on percent change from baseline in low-density lipoprotein cholesterol (LDL-C) in adults with heterozygous familial hypercholesterolemia (HeFH).

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 to ≤ 80 years of age
* Diagnosis of heterozygous familial hypercholesterolemia
* On a stable dose of an approved statin and lipid regulating medication
* Fasting LDL-C ≥ 100 mg/dL (2.6 mmol/L)
* Fasting triglycerides ≤ 400 mg/dL (4.5 mmol/L)

Exclusion Criteria:

* Homozygous familial hypercholesterolemia
* LDL or plasma apheresis
* New York Heart Association (NYHA) III or IV heart failure
* Uncontrolled cardiac arrhythmia
* Uncontrolled hypertension
* Type 1 diabetes, poorly controlled type 2 diabetes
* Uncontrolled hypothyroidism or hyperthyroidism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2013-02-07 (Actual); Primary Completion 2013-11-27 (Actual); Study Completion 2013-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (35):
- United States (2):
  - Research Site, Scottsdale, Arizona
  - Research Site, Cincinnati, Ohio
- Australia (2):
  - Research Site, Camperdown, New South Wales
  - Research Site, Perth, Western Australia
- Canada (4):
  - Research Site, Vancouver, British Columbia
  - Research Site, London, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Montreal, Quebec
- France (3):
  - Research Site, Bron
  - Research Site, Nantes
  - Research Site, Paris
- Research Site, Cologne, Germany
- Research Site, New Territories, Hong Kong
- Netherlands (7):
  - Research Site, Amersfoort
  - Research Site, Amsterdam
  - Research Site, Gouda
  - Research Site, Groningen
  - Research Site, Hoorn
  - Research Site, Tilburg
  - Research Site, Utrecht
- Research Site, Christchurch, New Zealand
- Research Site, Oslo, Norway
- South Africa (4):
  - Research Site, Johannesburg, Gauteng
  - Research Site, Midrand, Gauteng
  - Research Site, Observatory, Western Cape
  - Research Site, Parow, Western Cape
- Spain (4):
  - Research Site, Córdoba, Andalusia
  - Research Site, Zaragoza, Aragon
  - Research Site, Reus, Catalonia
  - Research Site, Madrid
- Research Site, Stockholm, Sweden
- Research Site, Reinach, Switzerland
- United Kingdom (3):
  - Research Site, Coventry
  - Research Site, London
  - Research Site, Manchester

REFERENCES:
- [Background] Toth PP, Descamps O, Genest J, Sattar N, Preiss D, Dent R, Djedjos C, Wu Y, Geller M, Uhart M, Somaratne R, Wasserman SM; PROFICIO Investigators. Pooled Safety Analysis of Evolocumab in Over 6000 Patients From Double-Blind and Open-Label Extension Studies. Circulation. 2017 May 9;135(19):1819-1831. doi: 10.1161/CIRCULATIONAHA.116.025233. Epub 2017 Mar 1. PMID 28249876
- [Background] Kuchimanchi M, Grover A, Emery MG, Somaratne R, Wasserman SM, Gibbs JP, Doshi S. Population pharmacokinetics and exposure-response modeling and simulation for evolocumab in healthy volunteers and patients with hypercholesterolemia. J Pharmacokinet Pharmacodyn. 2018 Jun;45(3):505-522. doi: 10.1007/s10928-018-9592-y. Epub 2018 May 7. PMID 29736889
- [Background] Kasichayanula S, Grover A, Emery MG, Gibbs MA, Somaratne R, Wasserman SM, Gibbs JP. Clinical Pharmacokinetics and Pharmacodynamics of Evolocumab, a PCSK9 Inhibitor. Clin Pharmacokinet. 2018 Jul;57(7):769-779. doi: 10.1007/s40262-017-0620-7. PMID 29353350
- [Background] Wasserman SM, Sabatine MS, Koren MJ, Giugliano RP, Legg JC, Emery MG, Doshi S, Liu T, Somaratne R, Gibbs JP. Comparison of LDL-C Reduction Using Different Evolocumab Doses and Intervals: Biological Insights and Treatment Implications. J Cardiovasc Pharmacol Ther. 2018 Sep;23(5):423-432. doi: 10.1177/1074248418774043. Epub 2018 May 16. PMID 29768954
- [Background] Raal FJ, Stein EA, Dufour R, Turner T, Civeira F, Burgess L, Langslet G, Scott R, Olsson AG, Sullivan D, Hovingh GK, Cariou B, Gouni-Berthold I, Somaratne R, Bridges I, Scott R, Wasserman SM, Gaudet D; RUTHERFORD-2 Investigators. PCSK9 inhibition with evolocumab (AMG 145) in heterozygous familial hypercholesterolaemia (RUTHERFORD-2): a randomised, double-blind, placebo-controlled trial. Lancet. 2015 Jan 24;385(9965):331-40. doi: 10.1016/S0140-6736(14)61399-4. Epub 2014 Oct 1. PMID 25282519
- [Background] Shapiro MD, Minnier J, Tavori H, Kassahun H, Flower A, Somaratne R, Fazio S. Relationship Between Low-Density Lipoprotein Cholesterol and Lipoprotein(a) Lowering in Response to PCSK9 Inhibition With Evolocumab. J Am Heart Assoc. 2019 Feb 19;8(4):e010932. doi: 10.1161/JAHA.118.010932. PMID 30755061
- [Background] Stroes E, Robinson JG, Raal FJ, Dufour R, Sullivan D, Kassahun H, Ma Y, Wasserman SM, Koren MJ. Consistent LDL-C response with evolocumab among patient subgroups in PROFICIO: A pooled analysis of 3146 patients from phase 3 studies. Clin Cardiol. 2018 Oct;41(10):1328-1335. doi: 10.1002/clc.23049. Epub 2018 Oct 21. PMID 30120772
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men and women 18 to 80 years old with a diagnosis of heterozygous familial hypercholesterolemia (HeFH) on stable doses of an approved statin with fasting low-density lipoprotein cholesterol (LDL-C) ≥ 100 mg/dL were eligible for this study. The first participant enrolled on 07 February 2013 and the last participant enrolled 03 September 2013.
Pre-assignment Details: Participants received subcutaneous placebo corresponding to the once monthly dose volume during a 6-week screening period. Those who completed the screening period and met final eligibility criteria were randomized 1:1:2:2 into 4 treatment groups. Randomization was stratified by LDL-C level (< 160 mg/dL vs ≥ 160 mg/dL) and ezetimibe use.
Period: Overall Study
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Started | 55 | 55 | 111 | 110
Received Treatment | 54 | 55 | 110 | 110
Completed | 49 | 54 | 101 | 108
Not Completed | 6 | 1 | 10 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 2
Not completed — Sponsor Decision | 4 | 0 | 9 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM | Total
Number analyzed (Participants) | 55 | 55 | 111 | 110 | 331
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (14.1) | 46.8 (12.1) | 52.3 (12.6) | 51.9 (12.0) | 51.1 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 45 | 46 | 140
  Male | 30 | 31 | 66 | 64 | 191
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 4 | 8 | 16
  Black or African American | 1 | 0 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 51 | 49 | 100 | 98 | 298
  Other | 2 | 3 | 6 | 3 | 14
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 54 | 55 | 111 | 109 | 329
Stratification Factor: Low-Density Lipoprotein Cholesterol (LDL-C) Level [Number; unit: participants]
  < 160 mg/dL | 35 | 35 | 70 | 70 | 210
  ≥ 160 mg/dL | 20 | 20 | 41 | 40 | 121
Baseline Ezetimibe Use [Number; unit: participants]
  No | 22 | 21 | 43 | 43 | 129
  Yes | 33 | 34 | 68 | 67 | 202
LDL-C Concentration [Mean (Standard Deviation); unit: mg/dL] — Data are provided for the full analysis set (all randomized participants who received at least
  1 dose of investigational product)
  mg/dL | 151.1 (36.5) | 151.5 (42.5) | 161.4 (51.0) | 153.6 (43.3) | 155.5 (44.9)
Non-High-Density Lipoprotein Cholesterol (non-HDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] — Data are provided for the full analysis set
  mg/dL | 175.4 (43.9) | 175.4 (45.9) | 187.4 (56.7) | 178.5 (45.8) | 180.4 (49.5)
Apolipoprotein B Concentration [Mean (Standard Deviation); unit: mg/dL] — Data are provided for the full analysis set
  mg/dL | 114.3 (29.8) | 110.3 (21.7) | 119.0 (30.7) | 114.9 (25.5) | 115.4 (27.5)
Total cholesterol/HDL-C Ratio [Mean (Standard Deviation); unit: ratio] — Data are provided for the full analysis set
  ratio | 4.695 (1.905) | 4.844 (1.435) | 5.159 (2.031) | 4.842 (1.801) | 4.924 (1.845)
Apolipoprotein B/Apolipoprotein A1 Ratio [Mean (Standard Deviation); unit: ratio] — Data are provided for the full analysis set
  ratio | 0.815 (0.264) | 0.851 (0.249) | 0.888 (0.322) | 0.850 (0.331) | 0.857 (0.305)
Lipoprotein(a) Concentration [Median (Inter-Quartile Range); unit: nmol/L] — Data are provided for the full analysis set
  nmol/L | 44.0 [24.0 to 105.0] | 87.0 [36.0 to 219.0] | 77.5 [29.0 to 205.5] | 61.0 [17.0 to 194.0] | 65.0 [25.0 to 199.0]
Triglyceride Concentration [Median (Inter-Quartile Range); unit: mg/dL] — Data are provided for the full analysis set
  mg/dL | 95.8 [74.5 to 143.0] | 102.0 [79.0 to 151.0] | 118.5 [86.5 to 160.5] | 112.5 [84.5 to 156.5] | 110.0 [81.5 to 154.0]
Very Low-Density Lipoprotein Cholesterol (VLDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] — Data are provided for the full analysis set
  mg/dL | 23.1 (10.7) | 23.9 (10.5) | 25.9 (11.8) | 24.9 (11.7) | 24.8 (11.4)
HDL-C Concentration [Mean (Standard Deviation); unit: mg/dL] — Data are provided for the full analysis set
  mg/dL | 53.2 (16.5) | 49.1 (12.7) | 50.4 (16.1) | 51.9 (16.0) | 51.1 (15.6)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in LDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set. Least squares (LS) means are from a repeated measures linear effects model; missing values were not imputed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 54 | 55 | 110 | 110
percent change | -2.02 (2.49) | 5.53 (3.25) | -61.25 (1.77) | -55.74 (2.25)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Within each dose frequency, the null hypothesis was that there was no mean difference in the percent change from baseline at week 12 or in the percent change from baseline at the mean of weeks 10 and 12 in LDL-C between evolocumab and placebo, and the alternative hypothesis was that a mean difference did exist; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The model includes treatment group, baseline LDL-C and ezetimibe use, scheduled visit, and the interaction of treatment with scheduled visit; LS Mean Treatment Difference = -59.23, 95% CI 2-sided [-65.11 to -53.35], Standard Error of Mean 2.98
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -61.27, 95% CI 2-sided [-69.00 to -53.55], Standard Error of Mean 3.91

2. Primary Outcome: Percent Change From Baseline in LDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 54 | 55 | 110 | 110
percent change | -1.08 (2.41) | 2.30 (2.41) | -61.23 (1.71) | -63.25 (1.70)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -60.15, 95% CI 2-sided [-65.83 to -54.46], Standard Error of Mean 2.88
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -65.55, 95% CI 2-sided [-71.27 to -59.83], Standard Error of Mean 2.90

3. Secondary Outcome: Change From Baseline in LDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 54 | 55 | 110 | 110
mg/dL | -6.5 (4.2) | -1.3 (4.1) | -101.7 (3.0) | -98.8 (2.9)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -95.2, 95% CI 2-sided [-105.1 to -85.2], Standard Error of Mean 5.0
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -97.4, 95% CI 2-sided [-107.1 to -87.7], Standard Error of Mean 4.9

4. Secondary Outcome: Change From Baseline in LDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 54 | 55 | 110 | 110
mg/dL | -8.5 (4.2) | 4.1 (5.2) | -101.3 (3.0) | -87.2 (3.6)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -92.9, 95% CI 2-sided [-102.9 to -82.8], Standard Error of Mean 5.1
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -91.3, 95% CI 2-sided [-103.8 to -78.9], Standard Error of Mean 6.3

5. Secondary Outcome: Percentage of Participants With Mean LDL-C at Weeks 10 and 12 of Less Than 70 mg/dL (1.8 mmol/L)
Time Frame: Weeks 10 and 12
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 54 | 55 | 110 | 110
percentage of participants | 1.9 [0.3 to 9.9] | 1.9 [0.3 to 9.8] | 67.0 [57.7 to 75.1] | 80.4 [71.9 to 86.8]
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Cochran-Mantel Haenszel test stratified by baseline LDL-C and ezetimibe use; Treatment Difference = 65.1, 95% CI 2-sided [52.8 to 73.4]
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Cochran-Mantel Haenszel test stratified by baseline LDL-C and ezetimibe use; Treatment Difference = 78.5, 95% CI 2-sided [66.9 to 85.1]

6. Secondary Outcome: Percentage of Participants With LDL-C < 70 mg/dL (1.8 mmol/L) at Week 12
Time Frame: Week 12
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 54 | 55 | 110 | 110
percentage of participants | 2.0 [0.3 to 10.3] | 2.2 [0.4 to 11.3] | 68.3 [58.8 to 76.4] | 63.1 [53.5 to 71.8]
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Cochran-Mantel Haenszel test stratified by baseline LDL-C and ezetimibe use; Treatment Difference = 66.3, 95% CI 2-sided [53.7 to 74.6]
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Cochran-Mantel Haenszel test stratified by baseline LDL-C and ezetimibe use; Treatment Difference = 60.9, 95% CI 2-sided [47.6 to 69.8]

7. Secondary Outcome: Percent Change From Baseline in Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 54 | 55 | 110 | 110
percent change | 0.21 (2.29) | 2.72 (2.21) | -55.79 (1.63) | -57.28 (1.56)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -56.00, 95% CI 2-sided [-61.41 to -50.59], Standard Error of Mean 2.74
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -60.01, 95% CI 2-sided [-65.24 to -54.77], Standard Error of Mean 2.65

8. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 54 | 55 | 110 | 110
percent change | -1.39 (2.40) | 5.29 (2.94) | -56.19 (1.71) | -49.67 (2.04)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -54.79, 95% CI 2-sided [-60.47 to -49.12], Standard Error of Mean 2.87
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -54.95, 95% CI 2-sided [-61.95 to -47.96], Standard Error of Mean 3.54

9. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 54 | 55 | 110 | 110
percent change | -0.19 (2.10) | 2.21 (1.97) | -49.58 (1.48) | -52.76 (1.36)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -49.39, 95% CI 2-sided [-54.32 to -44.46], Standard Error of Mean 2.50
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -54.98, 95% CI 2-sided [-59.58 to -50.38], Standard Error of Mean 2.33

10. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 54 | 55 | 110 | 110
percent change | -0.67 (2.32) | 4.60 (2.70) | -49.75 (1.63) | -44.81 (1.80)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -49.09, 95% CI 2-sided [-54.55 to -43.63], Standard Error of Mean 2.76
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -49.41, 95% CI 2-sided [-55.73 to -43.10], Standard Error of Mean 3.19

11. Secondary Outcome: Percent Change From Baseline in the Total Cholesterol/HDL-C Ratio at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 54 | 55 | 110 | 110
percent change | 0.86 (2.05) | 4.14 (2.13) | -45.74 (1.45) | -45.02 (1.50)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -46.59, 95% CI 2-sided [-51.43 to -41.76], Standard Error of Mean 2.45
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -49.16, 95% CI 2-sided [-54.21 to -44.11], Standard Error of Mean 2.56

12. Secondary Outcome: Percent Change From Baseline in the Total Cholesterol/HDL-C Ratio at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 54 | 55 | 110 | 110
percent change | 0.12 (2.19) | 7.11 (3.13) | -45.95 (1.56) | -38.32 (2.15)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -46.08, 95% CI 2-sided [-51.27 to -40.88], Standard Error of Mean 2.63
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -45.42, 95% CI 2-sided [-52.86 to -37.98], Standard Error of Mean 3.77

13. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B/Apolipoprotein A1 Ratio at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 54 | 55 | 110 | 110
percent change | 0.78 (2.21) | 1.65 (2.35) | -52.39 (1.56) | -53.91 (1.60)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -53.17, 95% CI 2-sided [-58.35 to -47.99], Standard Error of Mean 2.62
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -55.56, 95% CI 2-sided [-61.08 to -50.05], Standard Error of Mean 2.79

14. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B/Apolipoprotein A1 Ratio at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 54 | 55 | 110 | 110
percent change | 1.54 (2.49) | 4.23 (3.66) | -52.74 (1.75) | -45.31 (2.42)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -54.28, 95% CI 2-sided [-60.16 to -48.41], Standard Error of Mean 2.97
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -49.55, 95% CI 2-sided [-58.14 to -40.96], Standard Error of Mean 4.35

15. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 54 | 55 | 110 | 110
percent change | 7.34 (2.97) | 5.35 (2.95) | -24.03 (2.09) | -25.65 (2.07)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -31.37, 95% CI 2-sided [-38.33 to -24.41], Standard Error of Mean 3.52
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -31.00, 95% CI 2-sided [-37.91 to -24.09], Standard Error of Mean 3.50

16. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 54 | 55 | 110 | 110
percent change | 8.68 (3.27) | 6.69 (3.16) | -22.89 (2.31) | -21.55 (2.17)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -31.57, 95% CI 2-sided [-39.28 to -23.87], Standard Error of Mean 3.90
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -28.24, 95% CI 2-sided [-35.61 to -20.88], Standard Error of Mean 3.73

17. Secondary Outcome: Percent Change From Baseline in Triglycerides at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 54 | 55 | 110 | 110
percent change | 9.09 (3.02) | 7.49 (3.26) | -13.27 (2.14) | -9.25 (2.27)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -22.36, 95% CI 2-sided [-29.48 to -15.24], Standard Error of Mean 3.60
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -16.74, 95% CI 2-sided [-24.43 to -9.05], Standard Error of Mean 3.89

18. Secondary Outcome: Percent Change From Baseline in Triglycerides at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 54 | 55 | 110 | 110
percent change | 3.50 (3.51) | 6.43 (4.15) | -16.09 (2.49) | -5.13 (2.84)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -19.59, 95% CI 2-sided [-27.92 to -11.26], Standard Error of Mean 4.22
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -11.56, 95% CI 2-sided [-21.38 to -1.74], Standard Error of Mean 4.97

19. Secondary Outcome: Percent Change From Baseline in HDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 54 | 55 | 110 | 110
percent change | -0.45 (1.70) | -2.86 (1.84) | 7.93 (1.20) | 6.62 (1.29)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 8.38, 95% CI 2-sided [4.36 to 12.40], Standard Error of Mean 2.04
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 9.48, 95% CI 2-sided [5.10 to 13.85], Standard Error of Mean 2.21

20. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 54 | 55 | 110 | 110
percent change | -1.15 (1.91) | -3.73 (2.35) | 8.05 (1.35) | 5.35 (1.62)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 9.20, 95% CI 2-sided [4.66 to 13.74], Standard Error of Mean 2.30
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 9.07, 95% CI 2-sided [3.48 to 1466], Standard Error of Mean 2.83

21. Secondary Outcome: Percent Change From Baseline in Very Low-Density Lipoprotein Cholesterol (VLDL-C) at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 54 | 55 | 110 | 110
percent change | 8.66 (2.90) | 6.34 (3.27) | -13.97 (2.06) | -9.20 (2.27)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -22.63, 95% CI 2-sided [-29.46 to -15.81], Standard Error of Mean 3.46
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -15.54, 95% CI 2-sided [-23.25 to -7.84], Standard Error of Mean 3.90

22. Secondary Outcome: Percent Change From Baseline in VLDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 54 | 55 | 110 | 110
percent change | 3.73 (3.50) | 4.10 (4.17) | -17.25 (2.48) | -5.06 (2.84)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -20.97, 95% CI 2-sided [-29.29 to -12.66], Standard Error of Mean 4.21
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -9.17, 95% CI 2-sided [-19.01 to 0.68], Standard Error of Mean 4.98

ADVERSE EVENTS:
Time Frame: From the first dose of blinded investigational product until the end of the study (up to 14 weeks).
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Serious Adverse Events (participants affected / at risk) | 2/54 | 3/55 | 3/110 | 4/110
Other Adverse Events (participants affected / at risk) | 5/54 | 10/55 | 17/110 | 24/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=54) | Placebo QM (N=55) | Evolocumab Q2W (N=110) | Evolocumab QM (N=110)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0
Colonoscopy abnormal (Investigations) | 0 | 0 | 0 | 1
Endoscopy gastrointestinal abnormal (Investigations) | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=54) | Placebo QM (N=55) | Evolocumab Q2W (N=110) | Evolocumab QM (N=110)
Nasopharyngitis (Infections and infestations) | 2 | 3 | 8 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 7 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 6
Dizziness (Nervous system disorders) | 1 | 3 | 0 | 4
Headache (Nervous system disorders) | 1 | 3 | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.